CLINICAL TRIAL: NCT01172392
Title: A Randomized, Multicenter, Unblinded, Phase III Study Assessing the Loss of HbsAg at W96 After a 48-week Pegylated Interferon Alpha 2a in Patients With Chronic Hepatitis B (HbeAg Negative) Under Treatment and Responders (Undetectable Viral Load) to a Nucleoside(s) or Nucleotide(s) Analog(s) Treatment for at Least 12 Months. ANRS HB 06 Pegan
Brief Title: A Randomized Study to Assess the Loss of HbsAg After a 48-week Treatment Period With Pegylated Interferon Alpha 2a in Patients With Chronic Hepatitis B
Acronym: PEGAN
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010-019367-11; ANRS HB 06 PEGAN (Other: FrenchAIDS)
Record Dates: First submitted 2010-07-28; First posted 2010-07-29 (Estimated); Last update posted 2013-03-29 (Estimated); Status verified 2013-02

CONDITIONS: Chronic Hepatitis B; AgHbs Negativation
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — peginterferon alfa-2a

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PegIFN + Nucleosidic or Nucleotidic Analog (Experimental)
  Interventions: Drug: Pegylated interferon-alpha-2a
- Nucleosidic or Nucleotidic Analog (Active Comparator)
  Interventions: Drug: Nucleotidic or Nucleosidic Treatment

INTERVENTIONS:
Drug: Pegylated interferon-alpha-2a — 180 mcg / wk / SC from D0 to W48
  Arms: PegIFN + Nucleosidic or Nucleotidic Analog
Drug: Nucleotidic or Nucleosidic Treatment — Analog treatment according to investigators practice
  Arms: Nucleosidic or Nucleotidic Analog

SUMMARY:
The purpose of this study is to assess the loss of HbsAg after a 48-week pegylated interferon alpha 2a in patients with chronic hepatitis B (HBeAg negativation)

DETAILED DESCRIPTION:
The purpose of this study is to provide a therapeutical alternative to the use of an extended or undeterminated duration of treatment with prolonged nucleoside (s)/nucleotide (s)analog (s).

The duration of administration is not consensual, and in most cases followed by a virological relapse, so that, the prolonged use could lead to the occurrence of viral resistance and mutations.

It is therefore expected that treatment with pegylated interferon for 48 weeks in patients with undetectable HBV DNA by analog(s) may increase and promotes the loss of HbsAg and then promotes HbsAg seroconversion. In the absence of cirrhosis, the loss of HbsAg at 6 months would allow the end of treatment

ELIGIBILITY:
Inclusion Criteria:

* Positive Hbs Ag
* Negative HbeAg
* Plasma HBV DNA undetectable at pre-inclusion ever since 12 months
* ALT less than or equal to 5 times the upper limit of normal
* Non cirrhotic or Not Decompensated Cirrhosis (Child Pugh <7)
* Undetectable hepatocellular carcinoma in liver scan and / or alpha-fetoprotein rate <50 ng / ml
* Unchanged nucleoside (s) and / or nucleotide (s) treatment for at least three months (and not including telbivudine)
* Negative pregnancy test for childbearing women
* Signed informed consent
* Use of contraception for childbearing women

Exclusion Criteria:

* Polymorphonuclear neutrophils <1500/mm3
* Platelets <70.000/mm3
* Co-infections with HIV, HCV and / or HDV
* Prolonged excessive consumption of alcohol
* Active intravenous drug addiction
* Immunomodulators Treatment(eg interferons), ever since one year
* Immunosuppressive treatments terminated ever since one year
* Telbivudine treatment
* Long course steroid treatment (more than 4 weeks) by oral way
* History of severe epilepsy or current use of anticonvulsants
* Severe heart disease (eg heart failure stage III or IV NYHA class, myocardial infarction less than 6 months, ventricular arrhythmia requiring treatment, unstable angina or other significant cardiovascular disease)
* Chronic liver disease other than HBV-related (hemochromatosis, autoimmune hepatitis, metabolic liver disease, including Wilson's disease and a deficiency of alpha1-antitrypsin deficiency, alcoholic liver disease, exposure to toxins)
* Presence or suspicion of cancer or a history of cancer (except basal cell carcinoma or in situ carcinoma) within 5 years preceding the randomization
* Thyroid uncontrolled disease, abnormal TSH, elevated thyroid antibodies and clinical manifestations of thyroid dysfunction
* History of autoimmune disease (inflammatory digestive, idiopathic thrombocytopenic purpura, lupus erythematosus, autoimmune hemolytic anemia, scleroderma, severe psoriasis, rheumatoid arthritis ....) Or presence of autoantibodies at a significant rate
* Renal impairment (creatinine clearance <50 ml / min using the Cockroft formula), renal transplantation, hemodialysis
* Hypersensitivity to the active substance, interferon alpha or any component
* History of depression or psychiatric disorders and uncontrolled depression or uncontrolled psychiatric disorders
* Pregnancy or breastfeeding, or wish of pregnancy during the study period.
* Patients under legal protection or unable to express their consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2011-01; Primary Completion 2015-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
HbsAg negativation at week 96 | W96
  Percentage of patients with negative HbsAg at W96, i.e 12 months after a 48 weeks treatment with pegylated interferon

SECONDARY OUTCOMES:
Kinetics of HbsAg | W-6, W0, W12, W24 and W48
  Kinetics of HbsAg under treatment at W-6, W0, W12, W24 and W48 and after discontinuation of PegIFN alpha 2a at W72, W20 and W144

CONTACTS AND LOCATIONS:
Overall Officials: Marc BOURLIERE, MD, Study Chair — Hôpital Saint Joseph, Service d'hépatogastroentérologie, Marseille
Locations (1):
- Hôpital Saint Joseph, Service d'hépatogastroentérologie, Marseille, France

REFERENCES:
- [Derived] Bourliere M, Rabiega P, Ganne-Carrie N, Serfaty L, Marcellin P, Barthe Y, Thabut D, Guyader D, Hezode C, Picon M, Causse X, Leroy V, Bronowicki JP, Carrieri P, Riachi G, Rosa I, Attali P, Molina JM, Bacq Y, Tran A, Grange JD, Zoulim F, Fontaine H, Alric L, Bertucci I, Bouvier-Alias M, Carrat F; ANRS HB06 PEGAN Study Group. Effect on HBs antigen clearance of addition of pegylated interferon alfa-2a to nucleos(t)ide analogue therapy versus nucleos(t)ide analogue therapy alone in patients with HBe antigen-negative chronic hepatitis B and sustained undetectable plasma hepatitis B virus DNA: a randomised, controlled, open-label trial. Lancet Gastroenterol Hepatol. 2017 Mar;2(3):177-188. doi: 10.1016/S2468-1253(16)30189-3. Epub 2017 Jan 20. PMID 28404133
- See also: French National Agency for Research on AIDS and viral hepatitis website — http://www.anrs.fr